CLINICAL TRIAL: NCT03927417
Title: Influence of Ethnical Differences on the Oocyte Yield in Patients Undergoing IVF / ICSI Treatment in Different Countries
Brief Title: Influence of Ethnical Differences on the Egg Cell Collected in Patients Undergoing Fertility Treatment
Status: Completed | Type: Observational
Sponsor: ART Fertility Clinics LLC (Other)
Responsible Party: Principal Investigator, Barbara Lawrenz, Scientific Director, ART Fertility Clinics LLC
Other Study IDs: 1901-ABU-012-BL
Record Dates: First submitted 2019-04-23; First posted 2019-04-25 (Actual); Last update posted 2021-01-08 (Actual); Status verified 2021-01

CONDITIONS: Infertility
Keywords: oocyte yield; ethnicity; ovarian stimulation
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Investigators wants to analyze the differences considering the country of origin, ethnicity, characteristics, reproductive history and habits of participants undergoing in vitro fertilization (IVF) / intracytoplasmic sperm injection (ICSI) treatment as well as the stimulation outcome in regards to stimulation dosages and egg cell yield.

DETAILED DESCRIPTION:
Infertility is acknowledged worldwide as a major health concern with significant regional differences. The prevalence of infertility in women of reproductive age has been estimated to be one in every seven couples in the western world and one in every four couples in developing countries. Geographical, sociocultural / religious and ethnical dissimilarities contribute to these global variations in infertility prevalence. Infertility has a major impact on family stability in many cultures, especially in developing countries, where childlessness can impact sociocultural status.

So far, most fertility treatments are based on studies performed in Western countries and therefore mostly performed in Caucasian population and research regarding infertility causes and optimal treatments in other populations is scarce. The aim of this prospective study is therefore to analyze the differences in the basic parameters of the populations analyzed, considering the country of origin and ethnicity undergoing IVF/ICSI treatment as well as the stimulation outcome in regards to stimulation dosages and oocyte yield.

ELIGIBILITY:
Inclusion Criteria:

• Couples with primary / secondary infertility who are planned to undergo IVF / ICSI treatment in one of the above mentioned centers and who agree to take part in this study.

Exclusion Criteria:

* Couples planned for oocyte and sperm donation
* Couples in whom the female partner has a history of:
* Chemotherapy or radiation which impacts the ovarian reserve
* Surgery at the ovaries / adnex region
* Tubal ligation
* Reversal of tubal ligation
* Endometriosis
* Couples in whom the male partner has a history of:
* Chemotherapy / Radiation which impacts the semen result
* Surgery at the testicles
* Vasectomy
* Surgery for reversal of vasectomy

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Couples with primary / secondary infertility who are planned to undergo IVF / ICSI treatment
Sampling Method: Non-Probability Sample
Enrollment: 1117 (Actual)
Dates: Start 2019-04-30 (Actual); Primary Completion 2020-09-29 (Actual); Study Completion 2020-10-31 (Actual)

PRIMARY OUTCOMES:
Number of retrieved oocytes | 1 day
  Number of retrieved oocytes
Number of mature oocytes | 1 day
  Number of mature oocytes
Fertilization rate | 1 day
  Fertilization rate (% of fertilized oocytes per metaphase II oocytes injected in case of ICSI / per metaphase II oocytes inseminated in case of IVF)

CONTACTS AND LOCATIONS:
Overall Officials: Barbara Lawrenz, PhD, Principal Investigator — IVI RMA Abu Dhabi
Locations (1):
- IVI Middle East Fertility Clinic, Abu Dhabi, United Arab Emirates

REFERENCES:
- [Background] Inhorn MC, Patrizio P. Infertility around the globe: new thinking on gender, reproductive technologies and global movements in the 21st century. Hum Reprod Update. 2015 Jul-Aug;21(4):411-26. doi: 10.1093/humupd/dmv016. Epub 2015 Mar 22. PMID 25801630
- [Background] Niederberger C, Pellicer A, Cohen J, Gardner DK, Palermo GD, O'Neill CL, Chow S, Rosenwaks Z, Cobo A, Swain JE, Schoolcraft WB, Frydman R, Bishop LA, Aharon D, Gordon C, New E, Decherney A, Tan SL, Paulson RJ, Goldfarb JM, Brannstrom M, Donnez J, Silber S, Dolmans MM, Simpson JL, Handyside AH, Munne S, Eguizabal C, Montserrat N, Izpisua Belmonte JC, Trounson A, Simon C, Tulandi T, Giudice LC, Norman RJ, Hsueh AJ, Sun Y, Laufer N, Kochman R, Eldar-Geva T, Lunenfeld B, Ezcurra D, D'Hooghe T, Fauser BCJM, Tarlatzis BC, Meldrum DR, Casper RF, Fatemi HM, Devroey P, Galliano D, Wikland M, Sigman M, Schoor RA, Goldstein M, Lipshultz LI, Schlegel PN, Hussein A, Oates RD, Brannigan RE, Ross HE, Pennings G, Klock SC, Brown S, Van Steirteghem A, Rebar RW, LaBarbera AR. Forty years of IVF. Fertil Steril. 2018 Jul 15;110(2):185-324.e5. doi: 10.1016/j.fertnstert.2018.06.005. PMID 30053940
- [Background] Baker VL, Luke B, Brown MB, Alvero R, Frattarelli JL, Usadi R, Grainger DA, Armstrong AY. Multivariate analysis of factors affecting probability of pregnancy and live birth with in vitro fertilization: an analysis of the Society for Assisted Reproductive Technology Clinic Outcomes Reporting System. Fertil Steril. 2010 Sep;94(4):1410-1416. doi: 10.1016/j.fertnstert.2009.07.986. Epub 2009 Sep 9. PMID 19740463